CLINICAL TRIAL: NCT00544492
Title: Study of Pain, Anxiety, Complications Related to AV Fistula Cannulation in Chronic Hemodialysis Patients. A. Buttonhole vs. Rope Ladder Technique B. Catheters With Cylindrical Point vs. Catheters With Bevel Point in Rope Ladder Technique
Brief Title: Study of Pain, Anxiety and Complications Related to Cannulation of Arteriovenous (AV) Fistula in Chronic Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Bert Bammens, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S50619
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Dialysis; Fistula
Keywords: arteriovenous fistula; dialysis access; pain; anxiety; fistula related complications; aneurysm
MeSH Terms: conditions — Fistula; Arteriovenous Fistula; Pain; Anxiety Disorders; Aneurysm | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Experimental): Buttonhole cannulation technique
  Interventions: Device: catheter for AV fistula cannulation
- A2 (Active Comparator): Rope ladder cannulation technique
  Interventions: Device: catheter for AV fistula cannulation
- B1 (Experimental): Catheter with bevel point
  Interventions: Device: catheter for AV fistula cannulation
- B2 (Active Comparator): Catheter with cylindrical point
  Interventions: Device: catheter for AV fistula cannulation

INTERVENTIONS:
Device: catheter for AV fistula cannulation — catheters for buttonhole technique (blunt, bevel point), catheters for rope ladder technique (sharp, bevel point or sharp, cylindrical point)
  Other Names: Beldico 1425 cath; Beldico 1425 mf cath; Beldico 1425 mf cath blunt

SUMMARY:
A. Pain and other disadvantages of AV fistula cannulation can be limited by using the so-called buttonhole technique.

B. Till present in our center catheters with cylindrical points are used for cannulation of AV fistulas with the rope ladder technique. One can hypothesize that a catheter with a bevel point might have some advantages such as a larger entrance area and less traumatic cannulation. The latter may influence pain sensation of the patients.

The above background information gives rise to the following investigational questions:

A. Buttonhole vs rope ladder technique

1. Is pain sensation different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   AV fistula cannulation by buttonhole technique causes less pain than cannulation by rope ladder technique.
2. Is the level of anxiety different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   AV fistula cannulation by buttonhole technique causes less anxiety than cannulation by rope ladder technique.
3. Is bleeding time different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   Bleeding time is shorter when using buttonhole technique versus rope ladder technique.
4. Is the number and severity of complications related to AV fistula cannulation different between buttonhole and rope ladder technique?

   Hypothesis:

   When using the buttonhole technique for AV fistula cannulation the number and severity of complications is less than when using the rope ladder technique.

   B. Rope ladder technique using catheters with cylindrical vs. bevel point
5. Is pain sensation different when using rope ladder cannulation catheters with cylindrical as compared to bevel point?

Hypothesis:

AV fistula cannulation using bevel point catheters causes less pain than cannulation using cylindrical point catheters.

DETAILED DESCRIPTION:
A. Pain and other disadvantages of AV fistula cannulation can be limited by using the so-called buttonhole technique. It was described for the first time as the "contant site method" by Twardowski et al. The authors report on a patient in whom the fistula was too short to use the rope ladder technique. As an alternative, the access was cannulated at a "constant site". Later, in 1984, Krönung used the name "buttonhole puncture technique". It was used primarily in patients treated with home hemodialysis, where cannulation was performed by one single person (often by the patient himself). In order to form a perfect buttonhole it is indeed essential that the fistula is cannulated at exactly the same site and using exactly the same angle every single time. The buttonhole technique has been adopted by the recent "National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF K/DOQI) Guidelines" for vascular access. Studies show that patient pain scores and bleeding time after dialysis are positively influenced when using this cannulation technique.

B. Till present in our center catheters with cylindrical points are used for cannulation of AV fistulas with the rope ladder technique. One can hypothesize that a catheter with a bevel point might have some advantages such as a larger entrance area and less traumatic cannulation. The latter may influence pain sensation of the patients.

The above background information gives rise to the following investigational questions:

A. Buttonhole vs rope ladder technique

1. Is pain sensation different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   AV fistula cannulation by buttonhole technique causes less pain than cannulation by rope ladder technique.
2. Is the level of anxiety different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   AV fistula cannulation by buttonhole technique causes less anxiety than cannulation by rope ladder technique.
3. Is bleeding time different when using buttonhole cannulation as compared to rope ladder cannulation technique?

   Hypothesis:

   Bleeding time is shorter when using buttonhole technique versus rope ladder technique.
4. Is the number and severity of complications related to AV fistula cannulation different between buttonhole and rope ladder technique?

   Hypothesis:

   When using the buttonhole technique for AV fistula cannulation the number and severity of complications is less than when using the rope ladder technique.

   B. Ropeladder technique using catheters with cylindrical vs. bevel point
5. Is pain sensation different when using rope ladder cannulation catheters with cylindrical as compared to bevel point?

Hypothesis:

AV fistula cannulation using bevel point catheters causes less pain than cannulation using cylindrical point catheters.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis
* at least 18 years of age
* AV fistula for vascular access
* speaking the Dutch language

Exclusion Criteria:

* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
A. Buttonhole vs. rope ladder AV fistula cannulation, comparison of pain, anxiety, bleeding time and fistula related complications B. Rope ladder AV fistula cannulation using catheters with cylindrical vs. bevel point, comparison of pain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bert RM Bammens, MD, PhD, Principal Investigator — University Hospital Gasthuisberg Leuven, Belgium
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Sands JJ. Increasing AV fistulae and decreasing dialysis catheters: two aspects of improving patient outcomes. Blood Purif. 2007;25(1):99-102. doi: 10.1159/000096404. Epub 2006 Dec 14. PMID 17170544
- [Background] Allon M, Robbin ML. Increasing arteriovenous fistulas in hemodialysis patients: problems and solutions. Kidney Int. 2002 Oct;62(4):1109-24. doi: 10.1111/j.1523-1755.2002.kid551.x. PMID 12234281
- [Background] Marticorena RM, Hunter J, Macleod S, Petershofer E, Dacouris N, Donnelly S, Goldstein MB. The salvage of aneurysmal fistulae utilizing a modified buttonhole cannulation technique and multiple cannulators. Hemodial Int. 2006 Apr;10(2):193-200. doi: 10.1111/j.1542-4758.2006.00094.x. PMID 16623674
- [Background] Ball LK. The buttonhole technique for arteriovenous fistula cannulation. Nephrol Nurs J. 2006 May-Jun;33(3):299-304. PMID 16859201
- [Background] Lloyd G, McLauchlan A. Nurses' attitudes towards management of pain. Nurs Times. 1994 Oct 26-Nov 1;90(43):40-3. PMID 7984461
- [Background] McDonald DD, Sterling R. Acute pain reduction strategies used by well older adults. Int J Nurs Stud. 1998 Oct;35(5):265-70. doi: 10.1016/s0020-7489(98)00039-x. PMID 9839185
- [Background] Miller CD, Robbin ML, Allon M. Gender differences in outcomes of arteriovenous fistulas in hemodialysis patients. Kidney Int. 2003 Jan;63(1):346-52. doi: 10.1046/j.1523-1755.2003.00740.x. PMID 12472802
- [Background] The management of chronic pain in older persons: AGS Panel on Chronic Pain in Older Persons. American Geriatrics Society. J Am Geriatr Soc. 1998 May;46(5):635-51. doi: 10.1111/j.1532-5415.1998.tb01084.x. No abstract available. PMID 9588381